CLINICAL TRIAL: NCT07192094
Title: A Reinforced Mindfulness-Based Intervention to Reduce Problematic Drinking Among Hispanic Emerging Adults: Feasibility and Acceptability
Brief Title: A Reinforced Mindfulness-Based Intervention to Reduce Problematic Drinking Among Hispanic Emerging Adults
Acronym: Mindfulness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); UConn Health (Other)
Responsible Party: Principal Investigator, Michelle M. Hospital, PhD, LMHC, BBA, Associate Director, Community-Based Research Institute; Research Associate Professor, Department of Biostatistics; Community Engagement Core Leader, FIU-RCMI, Florida International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AA030976 (NIH); R01AA030976 (NIH)
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: MBSR; Young Adults; Heavy Episodic Drinking
Keywords: Young adults; College Students; Ages 18 - 25; Binge Drinking; Stress; Mindfulness; Stress Reduction; HRV; Contingency Management; MBSR; alcohol misuse
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Intervention Model Description: The RCT will include a total of 120 participants. Participants will be randomly assigned to either the active adapted Mindfulness-Based Stress Reduction intervention group (n=60) or to an assessment-only control group (n=60).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Sessions (Experimental): An adapted Mindfulness-Based Stress Reduction (MBSR) intervention group (n=60). The intervention is an adapted MBSR 8-week program (1.5 hour/week), and the sessions will be delivered by a facilitator on FIU MMC Campus. Participants will also complete 3 quantitative study assessments and undergo biomarker collections at 4 timepoints .
  Interventions: Behavioral: Mindfulness Sessions - 8 Week Program
- Assessments Only (No Intervention): Assessment-only control group (n=60). Participants randomly assigned to the control condition will not receive the mindfulness intervention but will complete all study assessments and biomarker collections at the same timepoints as the intervention group (i.e., baseline, post-intervention, 1-month follow-up, and biomarker collections at four timepoints). These participants will not attend any mindfulness group sessions but will be compensated for their participation in data collection activities.

INTERVENTIONS:
Behavioral: Mindfulness Sessions - 8 Week Program — A culturally, and developmentally adapted Mindfulness-Based Stress Reduction (MBSR) program for Hispanic (self-identified) emerging adult (EA) participants (ages 18-25 years old) over 8 weeks (1.5 hours/week).
  Arms: Mindfulness Sessions

SUMMARY:
This study is a trial to evaluate a mindfulness program designed for Hispanic young adults. Participants will be randomly assigned to one of two groups: (1) an in-person, 8-week mindfulness program (one 1.5-hour session per week at FIU's MMC campus), or (2) an assessment-only control group. Regardless of group assignment. Participants will be asked to complete online surveys at baseline, after an 8-week period, and again one month later. They will also be asked to provide a fingerpick blood sample and have their heart rate and blood pressure measured at four timepoints: baseline, 1 month, 2 months, and 3 months after baseline. Participation will involve up to 16 hours over approximately 14 weeks. This includes time for completing baseline assessments, participating in the 8-week intervention (if assigned), and completing post-program and follow-up assessments. There are no serious risks of participating in this study, but some of the questions during the assessments, interview, or the fingerpick may cause you discomfort. The main benefit from participating in this clinical trial is that participants may experience personal benefits from learning mindfulness techniques.

DETAILED DESCRIPTION:
The primary objective of this Randomized Control Trial (RCT) will be to maximize the ecological validity of a cultural, and developmental adaptation of the Mindfulness-Based Stress Reduction (MBSR) program for Hispanic (self-identified) emerging adult (EA) participants (ages 18-25 years old).

The study team will recruit individuals (n=120, 60 Intervention, 60 Control ) from the target population, Hispanic EA (18-25) all of whom will meet the following eligibility criteria: self-identified Hispanic, 18-25 years old, engaged in 2 or more occasions of heavy episodic drinking occasions (HED) (4/5 drinks in one sitting for females/males) during the previous 30-days, and are actively enrolled at FIU as a student.

The intervention will consist of eight weekly 1.5-hour group sessions led by a trained facilitator at FIU's MMC campus and participants will be randomly assigned (1:1 allocation) to either the active Mindfulness-Based Stress Reduction intervention group (n=60) or to an assessment-only control group (n=60).

Procedures for data collection, compensation, and biomarkers will be as follows: Participants who enroll in the full RCT will be compensated with gift cards for their time and effort in completing data collection activities at designated timepoints -. baseline, 1-month post-baseline, post-intervention (approximately 2 months post-baseline), and 1-month follow-up (approximately 3 months post-baseline).

Biomarker collection will include a fingerprick blood sample to test for the alcohol biomarker phosphatidylethanol (PEth), as well as assessments of heart rate variability (HRV) and blood pressure (BP) as physiological indicators of stress.

To enhance engagement and reinforce attendance, an evidence-based fixed escalating Contingency Management schedule will be implemented at the conclusion of each mindfulness session. The sessions will be recorded, transcribed, and coded for appropriate developmental and cultural content by the research team. The risks associated with participation are minimal, but can include discomfort from assessments, biomarker collections, and potential breach of confidentially but these are minimal and typical routine procedures. Anticipated benefits include participant enjoyment of the sessions, engagement in self-study, learning mindfulness techniques for managing stress, and potential positive outcomes from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Hispanic,
* 18-25 years old,
* engaged in 2 or more occasions of heavy episodic drinking occasions (HED) (4/5 drinks in one sitting for females/males) during the previous 30-days
* actively enrolled FIU student. Exclusion Criteria

Participants will be flagged for exclusion criteria if they report any of the following:

* Five or more binge drinking episodes (5+ drinks in one sitting) in the past 30 days, which averages more than once per week.
* Weekly or more frequent use of other substances, including non-prescribed prescription drugs, illegal drugs, inhalants, or synthetic drugs.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Post Intervention (within 1 week of completing the program)
  Acceptability of the program will be assessed at post-intervention using a study-developed survey consisting of Likert-scale items (1 = Strongly Disagree to 5 = Strongly Agree). The survey evaluates multiple domains, including appropriateness and relevance, ease of participation and feasibility, engagement and interest, perceived benefit, satisfaction, facilitator feedback, and acceptability of the companion rewards program. Higher scores indicate greater acceptability, and results will be summarized descriptively at the item and domain levels.
Feasibility - Retention | Post Intervention (within 1 week of completing the program) and follow-up (1-month post program completion)
  Retention will be assessed as the proportion of enrolled participants who complete the post- and follow-intervention assessments. Unit of measure: percentage of enrolled participants.
Feasibility - Attendance (intervention group only) | Baseline through Week 8 (end of intervention)
  Attendance will be assessed as the average number of sessions attended out of 8 total sessions. Unit of measure: mean number of sessions attended.

SECONDARY OUTCOMES:
Reduction in Heavy Episodic Drinking (PEth) | Baseline to Post Intervention (8 weeks), 1 month follow up (12 weeks)
  Change in levels of Phosphatidylethanol (PEth) from baseline to post-intervention and 1-month follow-up.
Reduction in alcohol consumption (self-report) | Baseline to Post Intervention (8 weeks), 1 month follow up (12 weeks)
  Change average number of drinking days
Change in Perceived Stress | Baseline to Post Intervention (8 weeks), 1 month follow up (12 weeks)
  Change in self reported stress using validated instruments in RedCap

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hospital, PhD, LMHC, Principal Investigator — Florida International University
Locations (1):
- Academic Health Center 5 (AHC 5), Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from the randomized clinical trial portion of the study (i.e., the Clinical Adaptation Trial) will be shared, not the formative research data. De-identified data will be submitted to the NIAAA Data Archive (NIAAADA) in accordance with NOT-AA-22-003. Shared data will include baseline, intervention, and follow-up assessment variables, as well as derived outcome measures.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be submitted to the NIAAA Data Archive semi-annually. Data will become available to the research community consistent with the NIAAADA sharing schedule and will remain available indefinitely.
Access Criteria: Qualified investigators may access the de-identified dataset through the NIAAA Data Archive. Investigators must obtain IRB approval at their own institution (and, if applicable, at FIU) and agree to the NIAAADA Data Use Terms and Conditions. For requests outside NIAAADA, data may be shared by the PI under a data-sharing agreement that prohibits participant re-identification, requires data destruction after analyses, restricts redistribution, and requires acknowledgment of the data source.
URL: https://nda.nih.gov/niaaa

REFERENCES:
- [Background] Hospital MM, Contreras-Perez ME, Alessi SM, Langwerden RJ, Morris SL, Wagner EF. Mindfulness as an early intervention for hazardous alcohol use among non-treatment seeking Latine emerging adults: A mini-review. Addict Behav. 2023 Oct;145:107759. doi: 10.1016/j.addbeh.2023.107759. Epub 2023 May 29. PMID 37276788